CLINICAL TRIAL: NCT00905814
Title: A Phase I Bioequivalence Study To Compare The Plasma Pharmacokinetics Of Five 1-mg And One 5-mg AG-013736 Tablets In Healthy Volunteers
Brief Title: A Bioequivalence Study Of AG-013736 Tablets In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: A4061052
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (BABA) (Other): Treatment A: One 5-mg FCIR tablet Treatment B: Five 1-mg FCIR tablets Subjects in this sequence will participate in 4 periods in the following order: B -> A -> B -> A
  Interventions: Drug: AG-013736
- Sequence 2 (ABAB) (Other): Treatment A: One 5-mg FCIR tablet Treatment B: Five 1-mg FCIR tablets Subjects in this sequence will participate in 4 periods in the following order: A -> B -> A -> B
  Interventions: Drug: AG-103736

INTERVENTIONS:
Drug: AG-013736 — single oral dose of film coated immediate release tablet (one 5-mg tablet for Treatment A and five 1-mg tablets for Treatment B)
  Other Names: axitinib
  Arms: Sequence 1 (BABA)
Drug: AG-103736 — single oral dose of film coated immediate release tablet (one 5-mg tablet for Treatment A and five 1-mg tablets for Treatment B)
  Other Names: axitinib
  Arms: Sequence 2 (ABAB)

SUMMARY:
The hypothesis of this study is that one 5 mg tablet of axitinib has similar drug concentrations in plasma compared to five 1 mg tablets of axitinib after oral dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 47 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram (ECG) and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* Evidence of significant disease of the blood, kidney, endocrine system, lungs, gastrointestinal, heart, liver, psychiatric, neurologic, or allergic (including drug allergies, but excluding season allergies).
* Active smokers or users of tobacco containing products and other drugs
* Pregnant or nursing females; females of childbearing potential including those with tubal ligation.

Ages: 21 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To establish bioequivalence of five 1 mg film coated immediate release (FCIR) tablets of AG-013736 to one 5 mg FCIR tablet of AG-013736. | 3 days per period

SECONDARY OUTCOMES:
To assess the safety and tolerability of single dose AG-013736 when administered as five 1 mg FCIR tablets and one 5 mg FCIR tablet. | 3 days per period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061052&StudyName=A%20Bioequivalence%20Study%20Of%20AG-013736%20Tablets%20%20In%20Healthy%20Volunteers